CLINICAL TRIAL: NCT02148796
Title: Randomized, Placebo-controlled, Multicenter Study to Assess the Efficacy, Safety and Tolerability of ORal Bacterial EXtract for the Prevention of Wheezing Lower Respiratory Tract Illness (ORBEX)
Brief Title: Oral Bacterial Extract for the Prevention of Wheezing Lower Respiratory Tract Illness
Acronym: ORBEX
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Arizona (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: ORBEX-BV2014/06
Record Dates: First submitted 2014-05-19; First posted 2014-05-28 (Estimated); Last update posted 2024-08-29 (Actual); Status verified 2024-08

CONDITIONS: Asthma; Wheezing
Keywords: Wheezing; Lower respiratory tract illness; Asthma; Atopy
MeSH Terms: conditions — Asthma; Respiratory Sounds | interventions — Broncho-Vaxom

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Broncho-Vaxom (BV) (Active Comparator): One capsule of Broncho-Vaxom for children contains: 3.5 mg of lyophilized bacterial lysates of Haemophilus influenzae, Streptococcus (pneumonia, pyogenes and sanguinis (viridans)), Klebsiella (pneumoniae and ozaenae), Staphylococcus aureus and Moraxella catarrhalis. The content of the capsule will be mixed with a palatable liquid such as fruit juice.
  Interventions: Drug: Broncho-Vaxom (BV)
- Placebo (Placebo Comparator): A placebo capsule will be used that will be indistinguishable from the active study drug.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Broncho-Vaxom (BV) — Active Ingredient: Lyophilised bacterial extract; Chemical Name: OM-85 BV; Strength: 3.5 mg; Excipients: bacterial extract, propyl gallate, sodium glutamate, mannitol, pregelatinised starch, magnesium stearate; Appearance: Blue and white capsule; Dosage Form: 3.5 mg capsule; Manufacturer: OM Pharma, Switzerland (OM stands for Omnia Medicamenta) Storage: Store in the original package
  Other Names: OM-85 BV VEGETAL; Broncho-Vaxom concentrate (bacterial lysate)
  Arms: Broncho-Vaxom (BV)
Other: Placebo — A placebo capsule will be used that will be indistinguishable from the active study drug.
  Arms: Placebo

SUMMARY:
The primary objective of this study is to evaluate if Broncho-Vaxom® given to high risk infants for 10 days, monthly, for two consecutive years can increase time to occurrence of the first episode of wheezing lower respiratory tract illness (WLRI) during a three year observation period off therapy.

DETAILED DESCRIPTION:
This is a five year parallel arm, double-blind, placebo-controlled trial for the prevention of WLRI into the third to seventh year of life (30 to 78 mo inclusive) in young children (6-18 months old) at increased risk for asthma. The trial will be divided into 2 periods. During the initial treatment period (first and second years in the study) participants will receive Broncho- Vaxom® (3.5 mg) or placebo for ten days each month for two consecutive years. This period will allow the observation of key secondary outcomes while participants are receiving therapy. The second period (third through fifth years in the study) will be a three year observation of the time to occurrence of the first WLRI episode (primary outcome) while off study drug along with the secondary outcomes noted above. During both the treatment and observation periods, participants will be managed by study physicians using a rescue algorithm applied in the PEAK trial commensurate with the NAEPP Expert Panel Report (EPR) III guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Adequate completion of informed consent process with written documentation. The participant's legally acceptable representative must have provided the appropriate written informed consent. Assent forms will not be used due to the age of the participant population; however, for procedures later in the study when participants are older, age appropriate assent will be obtained, if required by local Institutional Review Board (IRB).
* Age: 6-18 months of age inclusive at randomization which means 5 to 17 months of age inclusive on entry into the one month run-in period. At least half of all enrolled children will be between 6 and 12 months of age at randomization.
* Participants will meet at least one of the following criteria, which have been associated with an increased risk of wheezing respiratory illnesses and asthma: a) Parental history of asthma -or- b) Physician-diagnosed atopic dermatitis in the participant - or- c) Physician-diagnosed asthma in a blood sibling aged 4 years or more.
* Participants may be either male or female.
* Participants will have at least one parent/guardian who can communicate with the study staff to allow assessment of study outcomes. All study materials used by parent/guardian will be made available in English and in Spanish.

The child's parent/guardian must have a working direct contact telephone.

Exclusion Criteria:

* Participants may not have had more than two prior WLRI episodes.
* Participants may not have had any SWLRI episodes.
* Participants may not have a physician's diagnosis of asthma.
* Participants may not have a systemic illness (other than allergy) including (but not limited to) recurrent seizures, chronic gastroesophageal reflux (GER) requiring medical treatment, major congenital anomalies, physical and intellectual delay, cerebral palsy, chest surgery, tuberculosis or other chronic infections, primary or secondary immunodeficiency, gastrointestinal malformation or disease or cardiac disorder (except a hemodynamically insignificant atrial septal defect (ASD), ventricular septal defect (VSD) or benign heart murmur).
* Participants may not have been born earlier than 36 weeks of gestation.
* Participants may not have received oxygen for more than 5 days in the neonatal period, or received mechanical ventilation with the exclusion of ventilation during anesthesia for a minor surgical procedure.
* Participants may not have significant neurodevelopmental delay.
* Participants may not be below the 3rd percentile for weight.
* Participants may not have any other chronic lung disease; e.g. chronic lung disease of prematurity (CLDP) or cystic fibrosis.
* Participants may not have a history of any life-threatening respiratory illness that required intubation and mechanical ventilation.
* The participant's family may not be expected to relocate out of study area within 3 years of the initiation of the study.
* Participants may not have received inhaled or systemic corticosteroids for respiratory related illness ever, or for other conditions in the month prior to randomization.
* Participants may not have ever received immunotherapy.
* Participants may not have ever received i.v. gammaglobulins or systemic immunosuppressants.
* Participants may not have received probiotics (Lactobacilli and Bifidobacteria) in medicinal form; (i.e. not including food), regularly for more than 4 months in the 6 to <12 mo age group or 6 months in the 12 to 18 month group prior to enrollment.
* Participant has known sensitivity to any of the study products and any of the ingredients to be administered.
* Participant has previously been randomized in this study. Participants who failed run-in and were not randomized may have study participation terminated and then be re-enrolled for a second run-in period.
* Participant is currently enrolled in or has completed any other investigational device or drug study <30 days prior to screening, or is receiving other investigational agent(s).
* Participant has a significant medical condition(s), anticipated need for major surgery during the study, or any other kind of disorder that may be associated with increased risk to the participant, or may interfere with study assessments, outcomes, or the ability to provide written informed consent or comply with study procedures, in the Investigator's opinion.
* The one month run-in period will be used to evaluate adherence to study drug administration and electronic communication. At randomization the participant must continue to meet enrolment criteria and also have demonstrated 80% adherence to the placebo during treatment period; i.e. 8 out of 10 days and a75% response rate to weekly mobile phone text queries; i.e. 3 out of 4 weekly text queries.
* Ongoing infection (of any organ system) at the time of randomization. This includes infections that are being adequately treated.
* Unable or unlikely to complete study assessments or the study intervention poses undue risk to patient in the opinion of the Investigator.
* Families will speak English and/or Spanish.

Ages: 6 Months to 18 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 822 (Actual)
Dates: Start 2017-01-03 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
The time to the occurrence of the first WLRI episode in the observation period while not receiving study drug | ages 30 to 42 months at the end of treatment; ages 66 to 78 months at completion
  The time to the occurrence of the first WLRI episode in the observation period while not receiving study drug

SECONDARY OUTCOMES:
The time to first WLRI during the two treatment years while receiving study drug | ages 6 to 18 months at start of therapy; ages 30 to 42 months at completion
  The time to first WLRI during the two treatment years while receiving study drug
The annualized rate of WLRI episodes during the two years while receiving study drug | ages 6 to 18 months at start of therapy; ages 30 to 42 months at completion
  The annualized rate of WLRI episodes during the two years while receiving study drug
The annualized rate of WLRI episodes during the observation period while not receiving study drug | ages 30 to 42 months at the end of treatment; ages 66 to 78 months at completion
  The annualized rate of WLRI episodes during the observation period while not receiving study drug
The annualized rate of severe wheezing respiratory tract illness (SWLRI) episodes during the two treatment years while receiving study drug. | ages 6 to 18 months at start of therapy; ages 30 to 42 months at completion
  SWLRI episodes are defined as cough and wheezing > 24 hours AND any one of the following:
  * Use of more than 6 albuterol treatments in ≤48 hours.
  * Unscheduled care visit for acute wheezing in doctor's office, urgent care or emergency department -or- hospitalization for wheezing.
  * Use of systemic corticosteroid prescribed by a licensed medical provider for a wheezing illness with or without a clinical visit.
  * The annualized rate of SWLRI episodes during the two years while receiving study drug.
The annualized rate of severe wheezing respiratory tract illness (SWLRI) episodes during the observation period while not receiving study drug. | ages 30 to 42 months at the end of treatment; ages 66 to 78 months at completion
  The annualized rate of severe wheezing respiratory tract illness (SWLRI) episodes during the observation period while not receiving study drug.
Asthma at the end of the observation period | ages 30 to 42 months at the end of treatment; ages 66 to 78 months at completion
  Asthma at the end of the observation period defined by any of the following three elements:
  (a) a health care provider diagnosis of asthma with reports of: at least one episode of wheezing or asthma in the previous year or asthma controllers prescribed for at least 6 months during the previous year; or (b) >3 episodes of wheezing during the previous year 38 ("frequent wheezers"); or (c) any wheezing during the third observation year in children who wheezed during the first three years of life ("persistent wheezers").
Safety and tolerability of Broncho-Vaxom® while receiving study drug during the two year treatment period. | ages 6 to 18 months at start of therapy; ages 30 to 42 months at completion
  Safety and tolerability of Broncho-Vaxom® while receiving study drug during the two year treatment period
Safety and tolerability of Broncho-Vaxom® while receiving study drug during the observation period. | ages 30 to 42 months at the end of treatment; ages 66 to 78 months at completion
  Safety and tolerability of Broncho-Vaxom® while receiving study drug during the observation period, after study drug has been stopped.

OTHER OUTCOMES:
The proportion of episode free days (EFD) annualized for each year of study. | Treatment (2 yr) and observation periods
  shortness of breath, cough, chest retraction or tightness; 2) No unscheduled medical visits for respiratory symptoms AND 3) No use of any asthma medications, including albuterol before exercise.
Time to first systemic corticosteroid course | Treatment (2 yr) and observation periods
  Time to first systemic corticosteroid course
Number of systemic corticosteroid courses | Treatment (2 yr) and observation periods
  Number of systemic corticosteroid courses
Cumulative systemic corticosteroid courses | Treatment (2 yr) and observation periods
  Cumulative systemic corticosteroid courses
Cumulative systemic corticosteroid dose | Treatment (2 yr) and observation periods
  Cumulative systemic corticosteroid dose
Cumulative time receiving controller inhaled corticosteroid (ICS) | Treatment (2 yr) and observation periods
  Cumulative time receiving controller inhaled corticosteroid (ICS)
Cumulative does of controller ICS | Treatment (2 yr) and observation periods
  Cumulative does of controller ICS
Cumulative time of receiving any controller medication (ICS, systemic steroid, or montelukast) | Treatment (2 yr) and observation periods
  Cumulative time of receiving any controller medication (ICS, systemic steroid, or montelukast)
Days with albuterol use | Treatment (2 yr) and observation periods
  Days with albuterol use
Urgent care/Emergency Department (ED)/Office visits/hospitalizations for respiratory illness analyzed separately and combined variable | Treatment (2 yr) and observation periods
  Urgent care/ED/Office visits/hospitalizations for respiratory illness analyzed separately and combined variable
Change in height and weight from baseline | Treatment (2 yr) and observation periods
  Change in height and weight from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Fernando D Martinez, MD, Principal Investigator — University of Arizona; Wayne J Morgan, MD, Study Director — University of Arizona; Dave T Mauger, PhD, Study Director — Penn State University, Data Coordinating Center
Locations (11):
- United States (11):
  - Phoenix Children's Hospital, Phoenix, Arizona
  - University of Arizona, Tucson, Arizona
  - University of California San Francisco, Benioff Children's Hospital, Oakland, California
  - Children's National Health System, Washington D.C., District of Columbia
  - Emory University, Atlanta, Georgia
  - Boston Children's Hospital, Harvard University, Boston, Massachusetts
  - Washington University, St Louis, Missouri
  - Columbia University, New York, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Cincinnati Children's Hospital & Medical Center, Cincinnati, Ohio
  - University of Wisconsin, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ahanchian H, Jones CM, Chen YS, Sly PD. Respiratory viral infections in children with asthma: do they matter and can we prevent them? BMC Pediatr. 2012 Sep 13;12:147. doi: 10.1186/1471-2431-12-147. PMID 22974166
- [Background] Azad MB, Coneys JG, Kozyrskyj AL, Field CJ, Ramsey CD, Becker AB, Friesen C, Abou-Setta AM, Zarychanski R. Probiotic supplementation during pregnancy or infancy for the prevention of asthma and wheeze: systematic review and meta-analysis. BMJ. 2013 Dec 4;347:f6471. doi: 10.1136/bmj.f6471. PMID 24304677
- [Background] Becker A, Watson W, Ferguson A, Dimich-Ward H, Chan-Yeung M. The Canadian asthma primary prevention study: outcomes at 2 years of age. J Allergy Clin Immunol. 2004 Apr;113(4):650-6. doi: 10.1016/j.jaci.2004.01.754. PMID 15100668
- [Background] Beydon N, Davis SD, Lombardi E, Allen JL, Arets HG, Aurora P, Bisgaard H, Davis GM, Ducharme FM, Eigen H, Gappa M, Gaultier C, Gustafsson PM, Hall GL, Hantos Z, Healy MJ, Jones MH, Klug B, Lodrup Carlsen KC, McKenzie SA, Marchal F, Mayer OH, Merkus PJ, Morris MG, Oostveen E, Pillow JJ, Seddon PC, Silverman M, Sly PD, Stocks J, Tepper RS, Vilozni D, Wilson NM; American Thoracic Society/European Respiratory Society Working Group on Infant and Young Children Pulmonary Function Testing. An official American Thoracic Society/European Respiratory Society statement: pulmonary function testing in preschool children. Am J Respir Crit Care Med. 2007 Jun 15;175(12):1304-45. doi: 10.1164/rccm.200605-642ST. No abstract available. PMID 17545458
- [Background] Bisgaard H, Hermansen MN, Buchvald F, Loland L, Halkjaer LB, Bonnelykke K, Brasholt M, Heltberg A, Vissing NH, Thorsen SV, Stage M, Pipper CB. Childhood asthma after bacterial colonization of the airway in neonates. N Engl J Med. 2007 Oct 11;357(15):1487-95. doi: 10.1056/NEJMoa052632. PMID 17928596
- [Background] Bluestone JA, Auchincloss H, Nepom GT, Rotrosen D, St Clair EW, Turka LA. The Immune Tolerance Network at 10 years: tolerance research at the bedside. Nat Rev Immunol. 2010 Nov;10(11):797-803. doi: 10.1038/nri2869. PMID 20972473
- [Background] Bousquet J, Anto J, Auffray C, Akdis M, Cambon-Thomsen A, Keil T, Haahtela T, Lambrecht BN, Postma DS, Sunyer J, Valenta R, Akdis CA, Annesi-Maesano I, Arno A, Bachert C, Ballester F, Basagana X, Baumgartner U, Bindslev-Jensen C, Brunekreef B, Carlsen KH, Chatzi L, Crameri R, Eveno E, Forastiere F, Garcia-Aymerich J, Guerra S, Hammad H, Heinrich J, Hirsch D, Jacquemin B, Kauffmann F, Kerkhof M, Kogevinas M, Koppelman GH, Kowalski ML, Lau S, Lodrup-Carlsen KC, Lopez-Botet M, Lotvall J, Lupinek C, Maier D, Makela MJ, Martinez FD, Mestres J, Momas I, Nawijn MC, Neubauer A, Oddie S, Palkonen S, Pin I, Pison C, Rance F, Reitamo S, Rial-Sebbag E, Salapatas M, Siroux V, Smagghe D, Torrent M, Toskala E, van Cauwenberge P, van Oosterhout AJ, Varraso R, von Hertzen L, Wickman M, Wijmenga C, Worm M, Wright J, Zuberbier T. MeDALL (Mechanisms of the Development of ALLergy): an integrated approach from phenotypes to systems medicine. Allergy. 2011 May;66(5):596-604. doi: 10.1111/j.1398-9995.2010.02534.x. Epub 2011 Jan 24. PMID 21261657
- [Background] Carroll KN, Gebretsadik T, Griffin MR, Wu P, Dupont WD, Mitchel EF, Enriquez R, Hartert TV. Increasing burden and risk factors for bronchiolitis-related medical visits in infants enrolled in a state health care insurance plan. Pediatrics. 2008 Jul;122(1):58-64. doi: 10.1542/peds.2007-2087. PMID 18595987
- [Background] Castro-Rodriguez JA, Holberg CJ, Wright AL, Martinez FD. A clinical index to define risk of asthma in young children with recurrent wheezing. Am J Respir Crit Care Med. 2000 Oct;162(4 Pt 1):1403-6. doi: 10.1164/ajrccm.162.4.9912111. PMID 11029352
- [Background] Collet JP, Ducruet T, Kramer MS, Haggerty J, Floret D, Chomel JJ, Durr F. Stimulation of nonspecific immunity to reduce the risk of recurrent infections in children attending day-care centers. The Epicreche Research Group. Pediatr Infect Dis J. 1993 Aug;12(8):648-52. doi: 10.1097/00006454-199308000-00005. PMID 8414777
- [Background] Del-Rio-Navarro BE, Espinosa Rosales F, Flenady V, Sienra-Monge JJ. Immunostimulants for preventing respiratory tract infection in children. Cochrane Database Syst Rev. 2006 Oct 18;(4):CD004974. doi: 10.1002/14651858.CD004974.pub2. PMID 17054227
- [Background] De Prost Y - Clinical Study Report (BV-2002/1) Multicentric, randomized, double-blind, placebo-controlled study of the efficacy and safety of Broncho-Vaxom® (OM-85 BV) in children suffering from atopic dermatitis. - Clinical Study Report (30 January 2008).
- [Background] Ege MJ, Mayer M, Normand AC, Genuneit J, Cookson WO, Braun-Fahrlander C, Heederik D, Piarroux R, von Mutius E; GABRIELA Transregio 22 Study Group. Exposure to environmental microorganisms and childhood asthma. N Engl J Med. 2011 Feb 24;364(8):701-9. doi: 10.1056/NEJMoa1007302. PMID 21345099
- [Background] Evans SE, Scott BL, Clement CG, Larson DT, Kontoyiannis D, Lewis RE, Lasala PR, Pawlik J, Peterson JW, Chopra AK, Klimpel G, Bowden G, Hook M, Xu Y, Tuvim MJ, Dickey BF. Stimulated innate resistance of lung epithelium protects mice broadly against bacteria and fungi. Am J Respir Cell Mol Biol. 2010 Jan;42(1):40-50. doi: 10.1165/rcmb.2008-0260OC. Epub 2009 Mar 27. PMID 19329554
- [Background] FDA Center for Drug Evaluation and Research (CDER) - Orally Inhaled and Intranasal Corticosteroids: Evaluation of the Effects on Growth in Children. Guidance for Industry: March 2007.
- [Background] Fernandes RM, Bialy LM, Vandermeer B, Tjosvold L, Plint AC, Patel H, Johnson DW, Klassen TP, Hartling L. Glucocorticoids for acute viral bronchiolitis in infants and young children. Cochrane Database Syst Rev. 2013 Jun 4;2013(6):CD004878. doi: 10.1002/14651858.CD004878.pub4. PMID 23733383
- [Background] Gadomski AM, Brower M. Bronchodilators for bronchiolitis. Cochrane Database Syst Rev. 2010 Dec 8;(12):CD001266. doi: 10.1002/14651858.CD001266.pub2. PMID 21154348
- [Background] Guilbert TW, Morgan WJ, Krawiec M, Lemanske RF Jr, Sorkness C, Szefler SJ, Larsen G, Spahn JD, Zeiger RS, Heldt G, Strunk RC, Bacharier LB, Bloomberg GR, Chinchilli VM, Boehmer SJ, Mauger EA, Mauger DT, Taussig LM, Martinez FD; Prevention of Early Asthma in Kids Study,Childhood Asthma Research and Education Network. The Prevention of Early Asthma in Kids study: design, rationale and methods for the Childhood Asthma Research and Education network. Control Clin Trials. 2004 Jun;25(3):286-310. doi: 10.1016/j.cct.2004.03.002. PMID 15157730
- [Background] Guilbert TW, Morgan WJ, Zeiger RS, Mauger DT, Boehmer SJ, Szefler SJ, Bacharier LB, Lemanske RF Jr, Strunk RC, Allen DB, Bloomberg GR, Heldt G, Krawiec M, Larsen G, Liu AH, Chinchilli VM, Sorkness CA, Taussig LM, Martinez FD. Long-term inhaled corticosteroids in preschool children at high risk for asthma. N Engl J Med. 2006 May 11;354(19):1985-97. doi: 10.1056/NEJMoa051378. PMID 16687711
- [Background] Halterman JS, Aligne CA, Auinger P, McBride JT, Szilagyi PG. Inadequate therapy for asthma among children in the United States. Pediatrics. 2000 Jan;105(1 Pt 3):272-6. PMID 10617735
- [Background] Holt PG, Sly PD, Martinez FD, Weiss ST, Bjorksten B, von Mutius E, Wahn U. Drug development strategies for asthma: in search of a new paradigm. Nat Immunol. 2004 Jul;5(7):695-8. doi: 10.1038/ni0704-695. PMID 15224096
- [Background] Jackson DJ. The role of rhinovirus infections in the development of early childhood asthma. Curr Opin Allergy Clin Immunol. 2010 Apr;10(2):133-8. doi: 10.1097/ACI.0b013e3283352f7c. PMID 19996738
- [Background] Jackson DJ, Gangnon RE, Evans MD, Roberg KA, Anderson EL, Pappas TE, Printz MC, Lee WM, Shult PA, Reisdorf E, Carlson-Dakes KT, Salazar LP, DaSilva DF, Tisler CJ, Gern JE, Lemanske RF Jr. Wheezing rhinovirus illnesses in early life predict asthma development in high-risk children. Am J Respir Crit Care Med. 2008 Oct 1;178(7):667-72. doi: 10.1164/rccm.200802-309OC. Epub 2008 Jun 19. PMID 18565953
- [Background] Juniper EF, Guyatt GH, Feeny DH, Ferrie PJ, Griffith LE, Townsend M. Measuring quality of life in children with asthma. Qual Life Res. 1996 Feb;5(1):35-46. doi: 10.1007/BF00435967. PMID 8901365
- [Background] Klassen AF, Landgraf JM, Lee SK, Barer M, Raina P, Chan HW, Matthew D, Brabyn D. Health related quality of life in 3 and 4 year old children and their parents: preliminary findings about a new questionnaire. Health Qual Life Outcomes. 2003 Dec 22;1:81. doi: 10.1186/1477-7525-1-81. PMID 14690543
- [Background] Kusel MM, de Klerk NH, Kebadze T, Vohma V, Holt PG, Johnston SL, Sly PD. Early-life respiratory viral infections, atopic sensitization, and risk of subsequent development of persistent asthma. J Allergy Clin Immunol. 2007 May;119(5):1105-10. doi: 10.1016/j.jaci.2006.12.669. Epub 2007 Mar 13. PMID 17353039
- [Background] Lau S. What is new in the prevention of atopy and asthma? Curr Opin Allergy Clin Immunol. 2013 Apr;13(2):181-6. doi: 10.1097/ACI.0b013e32835eb7b1. PMID 23400030
- [Background] Maier RM, Palmer MW, Andersen GL, Halonen MJ, Josephson KC, Maier RS, Martinez FD, Neilson JW, Stern DA, Vercelli D, Wright AL. Environmental determinants of and impact on childhood asthma by the bacterial community in household dust. Appl Environ Microbiol. 2010 Apr;76(8):2663-7. doi: 10.1128/AEM.01665-09. Epub 2010 Feb 12. PMID 20154107
- [Background] Mansbach JM, Camargo CA Jr. Respiratory viruses in bronchiolitis and their link to recurrent wheezing and asthma. Clin Lab Med. 2009 Dec;29(4):741-55. doi: 10.1016/j.cll.2009.07.011. PMID 19892232
- [Background] Martinez FD. The connection between early life wheezing and subsequent asthma: The viral march. Allergol Immunopathol (Madr). 2009 Sep-Oct;37(5):249-51. doi: 10.1016/j.aller.2009.06.008. PMID 19875225
- [Background] Martinez FD. New insights into the natural history of asthma: primary prevention on the horizon. J Allergy Clin Immunol. 2011 Nov;128(5):939-45. doi: 10.1016/j.jaci.2011.09.020. PMID 22036094
- [Background] McMahon AW, Levenson MS, McEvoy BW, Mosholder AD, Murphy D. Age and risks of FDA-approved long-acting beta(2)-adrenergic receptor agonists. Pediatrics. 2011 Nov;128(5):e1147-54. doi: 10.1542/peds.2010-1720. Epub 2011 Oct 24. PMID 22025595
- [Background] Mitchell H, Senturia Y, Gergen P, Baker D, Joseph C, McNiff-Mortimer K, Wedner HJ, Crain E, Eggleston P, Evans R 3rd, Kattan M, Kercsmar C, Leickly F, Malveaux F, Smartt E, Weiss K. Design and methods of the National Cooperative Inner-City Asthma Study. Pediatr Pulmonol. 1997 Oct;24(4):237-52. doi: 10.1002/(sici)1099-0496(199710)24:43.0.co;2-h. PMID 9368258
- [Background] Morgan WJ, Crain EF, Gruchalla RS, O'Connor GT, Kattan M, Evans R 3rd, Stout J, Malindzak G, Smartt E, Plaut M, Walter M, Vaughn B, Mitchell H; Inner-City Asthma Study Group. Results of a home-based environmental intervention among urban children with asthma. N Engl J Med. 2004 Sep 9;351(11):1068-80. doi: 10.1056/NEJMoa032097. PMID 15356304
- [Background] Navarro RP, Schaecher KL, Rice GK. Asthma management guidelines: updates, advances, and new options. J Manag Care Pharm. 2007 Aug;13(6 Suppl D):S3-11; quiz S12-3. doi: 10.18553/jmcp.2007.13.s6-d.1. PMID 17713993
- [Background] Navarro S, Cossalter G, Chiavaroli C, Kanda A, Fleury S, Lazzari A, Cazareth J, Sparwasser T, Dombrowicz D, Glaichenhaus N, Julia V. The oral administration of bacterial extracts prevents asthma via the recruitment of regulatory T cells to the airways. Mucosal Immunol. 2011 Jan;4(1):53-65. doi: 10.1038/mi.2010.51. Epub 2010 Sep 1. PMID 20811345
- [Background] NHIS (2011)] National Health Interview Survey Data - Current Asthma Population Estimates. National Center for Health Statistics (NCHS), Centers for Disease Control and Prevention Hyattsville, MD: http://www.cdc.gov/asthma/nhis/2011/data.htm
- [Background] NHLBI. National Asthma Education and Prevention Program: Expert Panel Report 3: Guidelines for the Diagnosis and Management of Asthma; NIH Publication Number 08-5846. October 2007.
- [Background] Parola C, Salogni L, Vaira X, Scutera S, Somma P, Salvi V, Musso T, Tabbia G, Bardessono M, Pasquali C, Mantovani A, Sozzani S, Bosisio D. Selective activation of human dendritic cells by OM-85 through a NF-kB and MAPK dependent pathway. PLoS One. 2013 Dec 30;8(12):e82867. doi: 10.1371/journal.pone.0082867. eCollection 2013. PMID 24386121
- [Background] Principi N - Clinical Study Report (BV-2005/01) Double-Blind, Placebo-Controlled, Randomised Clinical Study of Broncho-Vaxom in Children Suffering from Recurrent Upper Respiratory Tract Infections. - Clinical Study Report (2 October 2012a).
- [Background] Pasquali C, Salami O, Taneja M, Gollwitzer ES, Trompette A, Pattaroni C, Yadava K, Bauer J, Marsland BJ. Enhanced Mucosal Antibody Production and Protection against Respiratory Infections Following an Orally Administered Bacterial Extract. Front Med (Lausanne). 2014 Oct 30;1:41. doi: 10.3389/fmed.2014.00041. eCollection 2014. PMID 25593914
- [Background] Principi N - Clinical Study Report (EBV09/01) Double-Blind, Placebo-Controlled, Randomised Clinical Study of Broncho-Vaxom® Drops in Children Suffering from Recurrent Respiratory Tract Infections. - Clinical Study Report (23 October 2012b).
- [Background] Razi CH, Harmanci K, Abaci A, Ozdemir O, Hizli S, Renda R, Keskin F. The immunostimulant OM-85 BV prevents wheezing attacks in preschool children. J Allergy Clin Immunol. 2010 Oct;126(4):763-9. doi: 10.1016/j.jaci.2010.07.038. PMID 20920766
- [Background] Riedler J, Braun-Fahrlander C, Eder W, Schreuer M, Waser M, Maisch S, Carr D, Schierl R, Nowak D, von Mutius E; ALEX Study Team. Exposure to farming in early life and development of asthma and allergy: a cross-sectional survey. Lancet. 2001 Oct 6;358(9288):1129-33. doi: 10.1016/S0140-6736(01)06252-3. PMID 11597666
- [Background] Schaad UB. OM-85 BV, an immunostimulant in pediatric recurrent respiratory tract infections: a systematic review. World J Pediatr. 2010 Feb;6(1):5-12. doi: 10.1007/s12519-010-0001-x. Epub 2010 Feb 9. PMID 20143206
- [Background] Sigurs N, Bjarnason R, Sigurbergsson F, Kjellman B. Respiratory syncytial virus bronchiolitis in infancy is an important risk factor for asthma and allergy at age 7. Am J Respir Crit Care Med. 2000 May;161(5):1501-7. doi: 10.1164/ajrccm.161.5.9906076. PMID 10806145
- [Background] Sly PD, Kusel M, Holt PG. Do early-life viral infections cause asthma? J Allergy Clin Immunol. 2010 Jun;125(6):1202-5. doi: 10.1016/j.jaci.2010.01.024. Epub 2010 Mar 20. PMID 20304476
- [Background] Spertini F - Clinical Study Report (BV-2007/03) Efficacy of Broncho-Vaxom® in Allergic Rhinitis: A Randomized, Double-Blind, Placebo-Controlled Phase IIa Study. - Clinical Study Report (31 July 2009)
- [Background] Strickland DH, Holt PG. T regulatory cells in childhood asthma. Trends Immunol. 2011 Sep;32(9):420-7. doi: 10.1016/j.it.2011.06.010. Epub 2011 Jul 27. PMID 21798806
- [Background] Strickland DH, Judd S, Thomas JA, Larcombe AN, Sly PD, Holt PG. Boosting airway T-regulatory cells by gastrointestinal stimulation as a strategy for asthma control. Mucosal Immunol. 2011 Jan;4(1):43-52. doi: 10.1038/mi.2010.43. Epub 2010 Jul 28. PMID 20668438
- [Background] Thorburn K, Harigopal S, Reddy V, Taylor N, van Saene HK. High incidence of pulmonary bacterial co-infection in children with severe respiratory syncytial virus (RSV) bronchiolitis. Thorax. 2006 Jul;61(7):611-5. doi: 10.1136/thx.2005.048397. Epub 2006 Mar 14. PMID 16537670
- [Background] Tuvim MJ, Evans SE, Clement CG, Dickey BF, Gilbert BE. Augmented lung inflammation protects against influenza A pneumonia. PLoS One. 2009;4(1):e4176. doi: 10.1371/journal.pone.0004176. Epub 2009 Jan 12. PMID 19137067
- [Background] von Mutius E, Vercelli D. Farm living: effects on childhood asthma and allergy. Nat Rev Immunol. 2010 Dec;10(12):861-8. doi: 10.1038/nri2871. Epub 2010 Nov 9. PMID 21060319
- [Background] Wildfire JJ, Gergen PJ, Sorkness CA, Mitchell HE, Calatroni A, Kattan M, Szefler SJ, Teach SJ, Bloomberg GR, Wood RA, Liu AH, Pongracic JA, Chmiel JF, Conroy K, Rivera-Sanchez Y, Busse WW, Morgan WJ. Development and validation of the Composite Asthma Severity Index--an outcome measure for use in children and adolescents. J Allergy Clin Immunol. 2012 Mar;129(3):694-701. doi: 10.1016/j.jaci.2011.12.962. Epub 2012 Jan 12. PMID 22244599
- [Background] Yasuda Y, Matsumura Y, Kasahara K, Ouji N, Sugiura S, Mikasa K, Kita E. Microbial exposure early in life regulates airway inflammation in mice after infection with Streptococcus pneumoniae with enhancement of local resistance. Am J Physiol Lung Cell Mol Physiol. 2010 Jan;298(1):L67-78. doi: 10.1152/ajplung.00193.2009. Epub 2009 Sep 25. PMID 19783640
- [Background] Yoo J, Tcheurekdjian H, Lynch SV, Cabana M, Boushey HA. Microbial manipulation of immune function for asthma prevention: inferences from clinical trials. Proc Am Thorac Soc. 2007 Jul;4(3):277-82. doi: 10.1513/pats.200702-033AW. PMID 17607013
- [Background] Yunginger JW, Reed CE, O'Connell EJ, Melton LJ 3rd, O'Fallon WM, Silverstein MD. A community-based study of the epidemiology of asthma. Incidence rates, 1964-1983. Am Rev Respir Dis. 1992 Oct;146(4):888-94. doi: 10.1164/ajrccm/146.4.888. PMID 1416415
- [Background] Zeiger RS, Mauger D, Bacharier LB, Guilbert TW, Martinez FD, Lemanske RF Jr, Strunk RC, Covar R, Szefler SJ, Boehmer S, Jackson DJ, Sorkness CA, Gern JE, Kelly HW, Friedman NJ, Mellon MH, Schatz M, Morgan WJ, Chinchilli VM, Raissy HH, Bade E, Malka-Rais J, Beigelman A, Taussig LM; CARE Network of the National Heart, Lung, and Blood Institute. Daily or intermittent budesonide in preschool children with recurrent wheezing. N Engl J Med. 2011 Nov 24;365(21):1990-2001. doi: 10.1056/NEJMoa1104647. PMID 22111718